CLINICAL TRIAL: NCT06043479
Title: Evaluation of the Effectiveness of the Training Given to Mothers With 0-5 Age Group Children for Fire Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Demet Yıldırım, nurse, Okan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Okan Uni
Record Dates: First submitted 2023-06-21; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Fever
Keywords: Child; fever,; mother,; fever management,; education
MeSH Terms: conditions — Fever

STUDY DESIGN:
Intervention Model Description: control group and intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The mothers were provided with a three-day training consisting of six sessions. Two sessions were held each day, with each session lasting for 30 minutes.
  Interventions: Other: Fever Management Education
- Control group (No Intervention): Routine practices continued for the mothers for three days without providing any training.

INTERVENTIONS:
Other: Fever Management Education — The mothers were provided with a three-day training consisting of six sessions. Two sessions were held each day, with each session lasting for 30 minutes.
  Arms: Intervention group

SUMMARY:
The research was conducted in a randomized controlled design to evaluate the effectiveness of the fever management training given to mothers of children aged 0-5.

DETAILED DESCRIPTION:
The research was conducted between January 2023 and April 2023 in the Pediatric Ward of Gebze Fatih State Hospital. The study included 120 mothers, with 60 in the intervention group and 60 in the control group, who had children aged 0-5 years old admitted to the hospital with a complaint of fever. The data was collected using the 'Mother and Child Information Form,' 'Parent's Fever Management Scale (PFMS),' 'Fever Management Knowledge Statements Form (FMKSF),' and 'Follow-up Form. The data were analyzed using appropriate statistical methods in the SPSS (Statistical Package for Social Sciences) for Windows 26.0 software package.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with 0-5 age group children in fever
* Must be literate

Exclusion Criteria:

* Discharge before 3 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Mother and Child Information Form | baseline
  The form was prepared by the researchers based on a literature review. It consists of 7 questions about the demographic characteristics of mothers and their children aged 0-5 years and mothers' fever management.
The Parent Fever Management Scale (PFMS) | baseline and 3 days and 1 month
  The scale was developed by Walsh and colleagues (2008), aims to assess what parents do when their child's temperature rises. Its validity and reliability have been established by Cinar et al. (2014). The scale consists of 8 items, and scores can range from 8 to 40. Higher scores on the scale indicate that parents engage in more fever management practices and have more concerns, fever phobia, and parental burden related to fever.
The Fever Management Knowledge Statements Form | baseline and 3 days and 1 month
  The form is a set of 25 statements developed by researchers to measure mothers' knowledge about fever management. These statements were created by reviewing the literature. Afterward, the statements were refined based on the input from five experts.
The Follow-up Form | through study completion, an average of 3 month
  The form was created by the researchers to track the participants' scores from the pre-test and post-test throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nadiye Barış Eren, Study Director — Tarsus University
Locations (1):
- .Demet Yildirim, Gebze, Kocaeli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No